CLINICAL TRIAL: NCT03395691
Title: Comparison of the Proximal Approach and Distal Approach of Axillary Vein Catheterization Under Ultrasound Guidance in Cardiac Surgical Patients With Risk of Bleeding: a Prospective Randomized Controlled Trial
Brief Title: Comparison of the Proximal Approach and Distal Approach of Axillary Vein Catheterization Under Ultrasound Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PANDA
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Central Venous Catheterization
Keywords: axillary vein; central venous catheterization; ultrasound; cardiac surgery; complication

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were randomized to the Proximal Approach (PA) or Distal Approach (DA) group in a 1:1 ratio using a computerized system. The allocation process was intensively managed by an allocation group using sequentially numbered containers and the allocation result was concealed until it was implemented. When a patient was eligible, the investigator informed allocation group to get intervention group allocated to the patient: PA or DA group. Because of feasibility issues, operators were not blinded to the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The distal approach (Active Comparator): The first two attempts via the distal approach will be performed . If the first two attempts failed, the subsequent attempts of venipuncture were performed using the proximal approach.
  Interventions: Procedure: The distal approach
- The proximal approach (Active Comparator): The first two attempts via the proximal approach will be performed . If the first two attempts failed, the subsequent attempts of venipuncture were performed using the distal approach.
  Interventions: Procedure: The proximal approach

INTERVENTIONS:
Procedure: The distal approach — The first two attempts via the distal approach will be performed . If the first two attempts failed, the subsequent attempts of venipuncture were performed using the proximal approach
  Arms: The distal approach
Procedure: The proximal approach — The first two attempts via the proximal approach will be performed . If the first two attempts failed, the subsequent attempts of venipuncture were performed using the distal approach.
  Arms: The proximal approach

SUMMARY:
Ultrasound-guided axillary vein catheterization can be performed via the proximal or distal approach of the axillary vein. The aim of our study is to compare the first puncture success rate and safety between the two approaches of ultrasound-guided axillary vein catheterization in cardiac surgical patients with risk of bleeding.

DETAILED DESCRIPTION:
For patients after cardiac surgery, antiplatelet drugs or anticoagulants are usually used for preventing thrombosis. Use of those drugs is associated with increased risk of bleeding. Any invasive procedures may put those patients at additional risk of bleeding. Ultrasound (US) has become widely accepted to guide safe and accurate central venous catheterization.The axillary vein in the infraclavicular area is an alternative choice for subclavian vein. Ultrasound images of the infraclavicular axillary vein differ according to its position. Proximal infraclavicular axillary vein is a direct continuation of the subclavian vein. The associated anatomy is simple and the vein is straight and thick in longitudinal axis view, which are in favor of successful puncture. Meanwhile, distal axillary vein also has anatomical advantages for safe and successful cannulations. Distal axillary vein lies further away from the artery and chest wall, and the overlap between distal axillary vein and artery gets greater on moving laterally. It is still unknow that one of the puncture approaches is superior to the other. Until now, there are no studies comparing two puncture approaches in high bleeding risk patients. The aim of the study is to compare the success rate of first puncture and safety of US-guided proximal and distal axillary venous catheterization in cardiac surgery patients with risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgical patients in Cardiac Surgery Intensive Care Unit
* Axillary vein catheterization is needed according to the clinical practice
* receiving oral antiplatelet or anticoagulants at least three days

Exclusion Criteria:

* fracture of the ipsilateral clavicle or anterior proximal ribs
* subclavian and/or axillary vein thrombosis
* local infection of the puncture area
* subclavian and/or axillary veins which are not clearly visualized using ultrasound
* already presence of subclavian or axillary vein catheter
* requiring an emergency axillary vein catheterization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-02-11 (Actual); Primary Completion 2019-09-14 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
First puncture success rate | approximately 3 minutes
  Central venous catheter established upon first punction attempt

SECONDARY OUTCOMES:
The approach success rate | within 1 hours
  the number of successful cannulation within the first two attempts
Complication rate | Day 1
  major bleeding, minor bleeding, arterial puncture, pneumothorax, nerve injuries, catheter misplacement
time to successful cannulation | within 1 hours
  the time from skin puncture until completion of cannula insertion
access time | within 1 hours
  defined as the time between penetration of skin and aspiration of venous blood into the syringe
overall success rate | within 1 hours
  defined as the number of successful cannulation in targeted axillary vein within four attempts (the first two attempts using the randomized approach, third and fourth attempts using the non-randomized approach)
the number of attempts | within 1 hours
  the number of attempts until successful cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Guo-wei Tu, PhD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buzancais G, Roger C, Bastide S, Jeannes P, Lefrant JY, Muller L. Comparison of two ultrasound guided approaches for axillary vein catheterization: a randomized controlled non-inferiority trial. Br J Anaesth. 2016 Feb;116(2):215-22. doi: 10.1093/bja/aev458. PMID 26787790
- [Background] Vezzani A, Manca T, Brusasco C, Santori G, Cantadori L, Ramelli A, Gonzi G, Nicolini F, Gherli T, Corradi F. A randomized clinical trial of ultrasound-guided infra-clavicular cannulation of the subclavian vein in cardiac surgical patients: short-axis versus long-axis approach. Intensive Care Med. 2017 Nov;43(11):1594-1601. doi: 10.1007/s00134-017-4756-6. Epub 2017 Mar 13. PMID 28289815
- [Derived] Su Y, Hou JY, Ma GG, Hao GW, Luo JC, Yu SJ, Liu K, Zheng JL, Xue Y, Luo Z, Tu GW. Comparison of the proximal and distal approaches for axillary vein catheterization under ultrasound guidance (PANDA) in cardiac surgery patients susceptible to bleeding: a randomized controlled trial. Ann Intensive Care. 2020 Jul 8;10(1):90. doi: 10.1186/s13613-020-00703-6. PMID 32643012